CLINICAL TRIAL: NCT02396706
Title: Randomized, Controlled, Double-blind, Multi-center Trial to Evaluate the Efficacy and Safety of a Liquid Containing Ivy Leaves Dry Extract vs. Placebo in the Treatment of Acute Cough
Brief Title: RCT to Evaluate the Efficacy and Safety of Ivy Leaves Cough Liquid vs. Placebo in the Treatment of Acute Cough
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Engelhard Arzneimittel GmbH & Co.KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EA-14-01-077
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Acute Cough

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Ivy Leaves Cough Liquid (Active Comparator): Ivy Leaves Cough Liquid
  Interventions: Drug: Ivy Leaves Cough Liquid
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivy Leaves Cough Liquid
  Arms: Ivy Leaves Cough Liquid
Drug: Placebo
  Arms: Placebo

SUMMARY:
Randomized, controlled, double-blind, multi-center trial to evaluate the efficacy and safety of a liquid containing ivy leaves dry extract vs. placebo in the treatment of acute cough

ELIGIBILITY:
Inclusion Criteria:

1. Acute cough with symptoms lasting 2-3 days prior to treatment
2. Men or women of any ethnic origin
3. Age 18 to 75 years
4. Subjects who are able to understand and are willing to comply to trial instructions
5. Having given written informed consent
6. Satisfactory health except for the cough as determined by the investigator based on medical history and physical examination
7. CS score of at least 50 mm on a 100 mm VAS at V1
8. Acute BSS of at least 10 points at V1
9. VCD score of at least 2 points at V1

Exclusion Criteria:

1. Allergic bronchial asthma, bronchial hyperreactivity, chronic bronchitis, other chronic or inherited lung disease
2. History of hypersensitivity to any excipient of the applied drugs
3. History of drug hypersensitivity, asthma, urticaria, or other severe allergic diathesis as well as current hay fever
4. History of chronic gastritis or peptic ulcers
5. Any gastrointestinal complaints within 7 days before V1
6. Participation in a clinical trial within 30 days prior to the treatment phase of this study or concomitantly
7. Treatment with corticoids, beta-2 agonists (e.g. salbutamol, fenoterol), expectorants, theophylline, antitussives, anaesthetics, acetylsalicylic acid (e.g. aspirin) or other non-steroidal anti-inflammatory drugs, leukotriene inhibitors, angiotensin-converting enzyme (ACE) inhibitors, antiviral drugs or antibiotics, antihistamines, immunosuppressants, isoprenaline, atropine, sodium cromoglycate or homeopathic drugs against common cold within 7 days before V1
8. Drug or alcohol abuse in the opinion of the investigator
9. Pregnant or nursing (lactating) women
10. Women of child-bearing potential (defined as all women physiologically capable of becoming pregnant) who are not using an acceptable method of contraception.
11. Subjects with significant diseases, defined as a disease which, in the opinion of the investigator, may either put the subject at risk because of participation in the trial or a disease which may influence the results of the trial or the subject's ability to participate in the trial; includes subjects with a history of gastrointestinal bleeding, significant cardiovascular, liver or renal disease.
12. Subjects directly or indirectly involved in the execution of this protocol, including employees of the CRO and persons related to them.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | whole treatment period over 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Axel Schaefer, Principal Investigator — Medizentrum Essen-Borbeck
Locations (1):
- Medizentrum Essen-Borbeck, Essen, Germany